CLINICAL TRIAL: NCT04998292
Title: Piezo-surgical Implant Placement With Laser
Brief Title: Piezo-surgical Implant With Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Sedky, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC/82-2021
Record Dates: First submitted 2021-07-19; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Effect of Piezo-surgical Implant With Laser on Pain and Swelling in Patients With Missing Teeth
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: split mouth study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy (Experimental)
  Interventions: Device: Piezo-surgery with low level laser therapy
- Control (Active Comparator)
  Interventions: Device: Piezo-surgery only

INTERVENTIONS:
Device: Piezo-surgery with low level laser therapy — Low level laser therapy
  Arms: Low level laser therapy
Device: Piezo-surgery only — Piezo-surgery only
  Arms: Control

SUMMARY:
Evaluation of the effect of laser with piezo-surgical device in dental implants

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects having good oral hygiene
* History of bilateral extractions in the lower molar area not less than 6 months ago.

Exclusion Criteria:

* Patients with debilitating diseases or bad oral hygiene,
* Patients with parafunctional habits and patients who are taking analgesics or with alcohol abuse.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-08-17 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain | 2 hours after surgery
Assessment of pain using visual analog scale | 6 hours after surgery
Assessment of pain using visual analog scale | 24 hours after surgery
Assessment of pain using visual analog scale | 2 days after surgery
Assessment of pain using visual analog scale | 3 days after surgery
Assessment of pain using visual analog scale | 4 days after surgery
Assessment of pain using visual analog scale | 7 days after surgery

SECONDARY OUTCOMES:
Swelling using swelling score system | 2 hours after surgery
Swelling using swelling score system | 6 hours after surgery
Swelling using swelling score system | 24 hours after surgery
Swelling using swelling score system | 2 days after surgery
Swelling | 3 days after surgery
Swelling using swelling score system | 4 days after surgery
Swelling using swelling score system | 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud, Cairo, Egypt